CLINICAL TRIAL: NCT04569357
Title: Multicenter Double-blind Placebo-controlled Parallel-group Randomized Clinical Trial of Efficacy and Safety of Prospekta in the Treatment of Attention Deficit/Hyperactivity Disorder in Children
Brief Title: Clinical Trial of Efficacy and Safety of Prospekta in the Treatment of Attention Deficit/Hyperactivity Disorder in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-MAP-004
Record Dates: First submitted 2020-09-22; First posted 2020-09-29 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2021-11

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: in children
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: double-blind placebo-controlled randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prospekta (Experimental): One tablet per intake 2 times a day (approximately at the same time), outside of meal (between meals or 15 minutes prior to meal or drinking). The tablet should be held in mouth until completely dissolved.
  Interventions: Drug: Prospekta
- Placebo (Placebo Comparator): One tablet per intake 2 times a day (approximately at the same time), outside of meal (between meals or 15 minutes prior to meal or drinking). The tablet should be held in mouth until completely dissolved.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prospekta — Oral administration.
  Other Names: MMH-MAP
  Arms: Prospekta
Drug: Placebo — Oral administration.
  Arms: Placebo

SUMMARY:
Purpose of the study:

• evaluate the efficacy and safety of Prospekta in the treatment of attention deficit/hyperactivity disorder in children.

DETAILED DESCRIPTION:
Design: a multicenter double-blind placebo-controlled parallel-group randomized clinical trial.

The study will enroll children of either age from 7 to 12 years old with diagnosis of attention deficit/hyperactivity disorder (ADHD) verified by Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, American Psychiatric Association" [DSM-V]).

After signing patient information sheet and informed consent form by the subject's parent/adoptive parent collection of complaints, medical examination of the children, filling Attention Deficit Hyperactivity Disorder-Rating Scale-V [ADHD-RS-V]) scale by the parent/adoptive parent will be performed, concomitant therapy will be recorded and laboratory tests will be carried out.

The study will enroll children with total score ADHD-RS-V ≥ 22. If the inclusion criteria were met and there were no exclusion criteria (Day 1), the patient will be randomized to one of the two groups: group 1 will receive Prospekta at 1 tablet twice daily; group 2 will receive Placebo using the study drug dosing regimen.

Treatment period will be 8 weeks, the key examination stages (collection of complaints, recording objective examination findings, repeated filling ADHD-RS-V by parent/adoptive parent) will be made at Visit 1 (Day 1), further in 4 weeks (visit 2) and in 8 weeks (visit 3). Each visit to the research center will be made by the subject accompanied by his/her parent/adoptive parent. Two weeks later (visit 1.1, week 2±3 days) after randomization and initiation of the study therapy and between visits 2 and 3 (visits 2.2, week 6±3 days) the investigator will examine the patient's clinical status (during phone calls). Based on complaints, monitoring of the prescribed therapy therapeutic safety will be assessed. At visit 2 (week 4±3 days) and visit 3 (week 8±3 days) the investigator will collect complaints, record objective examination findings, monitor repeated ADHD-RS-V filling by parent/adoptive parent, the prescribed and concomitant therapy, evaluate therapeutic safety and compliance. In addition at Visit 3 the investigator will complete the Clinical Global Impression Efficacy Index [CGI-EI] scale and collect samples for laboratory testing. The study treatments will be completed.

The total length of the observation period is 8 weeks. During the study the treatment for underlying conditions will be allowed with the exception of the drugs indicated in the section "Prohibited concomitant therapy".

ELIGIBILITY:
Inclusion Criteria:

1. Male and female children aged 7-12 years old inclusive.
2. Children with verified diagnosis of ADHD.
3. Presence of all ADHD criteria according to DSM-V (see appendix 1):

A. persistent pattern of inattention and/or hyperactivity-impulsivity that interferes with functioning or development, as characterized by (1) and/or (2):

1. Attention deficit: Six (or more) of the following symptoms have persisted for at least 6 months to a degree that is inconsistent with developmental level and that negatively impacts directly on social and academic/occupational activities:

   * Often fails to give close attention to details or makes careless mistakes in schoolwork, at work, or during other activities (e.g., overlooks or misses details, work is inaccurate).
   * Often has difficulty sustaining attention in tasks or play activities (e.g., has difficulty remaining focused during lectures, conversations, or lengthy reading).
   * Often does not seem to listen when spoken to directly (e.g., mind seems elsewhere, even in the absence of any obvious distraction).
   * Often does not follow through on instructions and fails to finish schoolwork, chores, or duties in the workplace (e.g., starts tasks but quickly loses focus and is easily sidetracked).
   * Often has difficulty organizing tasks and activities (e.g., difficulty managing sequential tasks; difficulty keeping materials and belongings in order; messy, disorganized work; has poor time management; fails to meet deadlines).
   * Often avoids, dislikes, or is reluctant to engage in tasks that require sustained mental effort (e.g., schoolwork or homework).
   * Often loses things necessary for tasks or activities (e.g., school materials, pencils, books, tools, wallets, keys, eyeglasses).
   * Is often easily distracted by extraneous stimuli.
   * Is often forgetful in daily activities (e.g., doing chores, running errands).
2. Hyperactivity/impulsivity: Six (or more) of the following symptoms have persisted for at least 6 months to a degree that is inconsistent with developmental level and that negatively impacts directly on social and academic/occupational activities. Note. The symptoms are not solely a manifestation of oppositional behavior, defiance, hostility, or failure to understand tasks or instructions.

   * Often fidgets with or taps hands or feet or squirms in seat.
   * Often leaves seat in situations when remaining seated is expected (e.g., leaves his or her place in the classroom, in the office or other workplace, or in other situations that require remaining in place).
   * Often runs about or climbs in situations where it is inappropriate.
   * Often unable to play or take part in leisure activities quietly.
   * Is often "on the go" acting as if "driven by a motor" (e.g., is unable to be or uncomfortable being still for extended time).
   * Often talks excessively.
   * Often blurts out an answer before a question has been completed (e.g., completes people's sentences; cannot wait for turn in conversation).
   * Often has trouble waiting his/her turn (e.g., while waiting in line).
   * Often interrupts or intrudes on others (e.g., butts into conversations, games, or activities; may start using other people's things without asking or receiving permission).

B. Several inattentive or hyperactive-impulsive symptoms were present before age 12 years.

C. Several inattentive or hyperactive-impulsive symptoms are present in two or more settings, (e.g., at home, school or work; with friends or relatives).

D. There is clear evidence that the symptoms interfere with, or reduce the quality of, social, school, or work functioning.

E. The symptoms do not occur exclusively during the course of schizophrenia or another psychotic disorder and are not better explained by another mental disorder (e.g., mood disorder, anxiety disorder, dissociative disorder, personality disorder, substance intoxication or withdrawal).

4. ADHD-RS-V ≥ 22. 5. Availability of signed information sheet and informed consent form for the parents/adoptive parents for the subject's participation in the clinical trial.

Exclusion Criteria:

1. History of central nervous system (CNS) diseases including:

   * Inflammatory diseases of the central nervous system (G00-G09).
   * Systemic atrophies primarily affecting the CNS (G10-G13).
   * Extrapyramidal and movement disorders (G20-G26).
   * Other degenerative diseases of the nervous system (G30-G32).
   * Demyelinating diseases of the CNS (G35-G37).
   * Epilepsy (G40-41).
   * Hydrocephalus (G91).
2. Childhood autism (F84.0), atypical autism • (F84.1).
3. Mental retardation (F70-79).
4. Disorders of psychological development (F80-F89).
5. History of hyperthyroidism (thyrotoxicosis).
6. History/suspicion of oncology of any location (except for benign neoplasms).
7. Any other comorbidity which, in the opinion of the investigator, may affect patient participation in the clinical trial.
8. Patients allergic to/intolerant of any constituent of the medications used in the treatment.
9. Hereditary lactose intolerance, malabsorption due to lactose intolerance including congenital or acquired lactase (or other disaccharide) deficiency, galactosemia.
10. Patients whose parents/adoptive parents will not fulfill the requirements during the study or follow the order of administration of the study drug (SD) products, from the Investigator's point of view.
11. History of treatment noncompliance, mental diseases, alcoholism or drug abuse in parents/adoptive parents which, according to the investigator, will prevent from following the study procedures.
12. Administration of the products outlined in section "Prohibited concomitant therapy" within 1 month prior to enrollment.
13. Patients who have participated in other clinical trials in the past 3 months.
14. The patient's parent/adoptive parent is a study specialist of the center and is directly involved in the study, or is an immediate family member of the Investigator. Spouses, parents, children, or siblings, regardless of whether they are siblings or adopted are considered immediate family members.
15. The patient's parent/adoptive parent works at Materia Medica Holding, i.e. they are employees of the Company, temporary employees on a contract basis or appointed officials responsible for conduction of the study or their immediate family members.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 363 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- Russia (31):
  - Hospital "Russian Railways - Medicine" of the city of Bryansk, Bryansk
  - Regional Clinical Specialized Psychoneurological Hospital # 1/Children's dispensary department, Chelyabinsk
  - Engels Psychiatric Hospital, Engel's
  - Kazan State Medical University/Department of Neurology, Neurosurgery and Medical Genetics, Kazan'
  - Children's Republican Clinical Hospital/Neurological department for the treatment of patients with CNS lesions with mental disorders, Kazan'
  - Specialized Clinical Psychiatric Hospital # 1/Dispensary department, Krasnodar
  - Russian National Research Medical University named after N.I. Pirogov/Department of Neurology, Neurosurgery and Medical Genetics, Faculty of Pediatrics, Moscow
  - Research and Practical Center of Pediatric Psychoneurology of Moscow City Health Department/Consultative and polyclinic department, Moscow
  - Moscow Regional Research Clinical Institute named after M.F. Vladimirsky/Neurology Department of Therapy Department, Moscow
  - Llc "Nizhmedklinika", Nizhny Novgorod
  - Privolzhsky Research Medical University/Department of Neurology, Psychiatry and Narcology FDPO, Nizhny Novgorod
  - Orenburg Regional Clinical Psychiatric Hospital # 1/Children's psychiatric department, Orenburg
  - Perm State Medical University named after academician E.A. Wagner/Department of Neurology, Perm
  - LLC "Treatment and rehabilitation research center "PHOENIX"/Day hospital # 1, Rostov-on-Don
  - Ryazan State Medical University named after Acad. I.P. Pavlov/Department of Children's Diseases with a course of hospital pediatrics, Ryazan
  - National Medical Research Center for Psychiatry and Neurology named after V.M. Bekhterev, Saint Petersburg
  - Llc "Doctrina", Saint Petersburg
  - Institute of the Human Brain named after N.P. Bekhtereva, Saint Petersburg
  - LLC "DNA Research Center", Saratov
  - Saratov State Medical University named after V.I. Razumovsky/Department of Neurology. named after K.N. Tretyakov, Saratov
  - City Clinical Hospital # 2 named after V.I. Razumovsky, Saratov
  - Saratov City Psychoneurological Dispensary, Saratov
  - Smolensk Regional Clinical Hospital/Children's neurological department, Smolensk
  - Smolensk Regional Clinical Hospital/Pediatric neurological department, Smolensk
  - LLC "Sunterra", Stavropol
  - Stavropol Regional Clinical Specialized Psychiatric Hospital # 1/Children's department # 17, Stavropol
  - Regional Clinical Psychoneurological Dispensary/Outpatient clinic # 2, Tver'
  - Children's City Clinical Hospital of Ulyanovsk city, Ulyanovsk
  - Yaroslavl State Medical University/Department of Polyclinic Pediatrics, Yaroslavl
  - Sverdlovsk Regional Clinical Psychiatric Hospital/Pediatric and adolescent medical and diagnostic department, Yekaterinburg
  - LLC "European Medical Center "UMMC-Health"/Children's polyclinic in the main branch, Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prospekta | Placebo
Started | 174 | 189
Completed | 174 | 189
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prospekta | Placebo | Total
Number analyzed (Participants) | 174 | 189 | 363
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 174 | 189 | 363
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.3 (1.7) | 9.3 (1.7) | 9.3 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 66 | 130
  Male | 110 | 123 | 233
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 174 | 189 | 363

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Total ADHD-RS-V Reduction ≥25%
Description: Attention Deficit Hyperactivity Disorder-Rating Scale-V (ADHD-V). The home version of ADHD-RS-V will be used separately for children (7-10 years old) and teenagers (11-12 years old). Home version will evaluate behaviour and emotional response in the situations in which the child is with his/her parents. ADHD-RS-V will evaluate 18 symptoms presented as brief characteristics of peculiarities in behaviour and emotional response of children in various situations (at home).
Time Frame: After 8 weeks of treatment
Population: There is no data on the ADHD-RS-V questionnaire after 8 weeks of treatment from 4 patients in the Prospekta group and 2 patients in the Placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 170 | 187
Participants | 95 | 81
Statistical Analysis 1: Comparison: Prospekta vs Placebo; Test for comparison percentage of patients with reduction ≥ 25%; Test type: Superiority; p = 0.0199, Fisher Exact

2. Secondary Outcome: Change in Total Attention Deficit Hyperactivity Disorder-Rating Scale-V (ADHD-RS-V) Score
Description: Attention Deficit Hyperactivity Disorder-Rating Scale-V (ADHD-RS-V). Versus baseline. The home version of ADHD-RS-V will be used separately for children (7-10 years old) and teenagers (11-12 years old). The home version of ADHD-RS-V will evaluate 18 symptoms presented as brief characteristics of peculiarities in behaviour and emotional response of children in various situations (at home, with his/her parents). The home version of ADHD-RS-V includes two subscales, one for attention deficit and one for hyperactivity-impulsivity. Each item is responded to using a four-point Likert scale, where 0 - "never or rarely"; 1 - "sometimes"; 2 - "often"; 3 - "very often." Total score for scale is to be formed using summations of all items. The maximum possible number of points is 54. The minimum score is 0. Higher score = more severe ADHD symptoms.
Time Frame: After 8 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 170 | 187
score on a scale
  Baseline | 32.5 (6.0) | 32.7 (6.3)
  After 4 weeks of treatment | 27.6 (6.2) | 28.2 (6.4)
  After 8 weeks of treatment | 22.3 (7.4) | 24.6 (8.7)
  ∆ between baseline and after 8 weeks of treatment | 10.2 (7.7) | 8.1 (7.9)
Statistical Analysis 1: Comparison: Prospekta vs Placebo; Mean changes of ADHD-RS-V scores after 8 weeks of treatment were compared; Test type: Superiority; p = 0.0096, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Total ADHD-RS-V Attention Deficit Subscale Score
Description: Attention Deficit Hyperactivity Disorder-Rating Scale-V (ADHD-RS-V). Attention deficit subscale. Versus baseline. The home version of ADHD-RS-V will be used separately for children (7-10 years old) and teenagers (11-12 years old). The home version of ADHD-RS-V includes two subscales, one for attention deficit and one for hyperactivity/impulsivity. The attention deficit items are: (1) Attention to detail; (2) Sustaining attention; (3) Does not seem to listen; (4) Follows instructions; (5) Difficulty organizing; (6) Sustained mental effort; (7) Loses things; (8) Distracted; (9) Forgetful. Each item is responded to using a four-point Likert scale, where 0 - "never or rarely"; 1 - "sometimes"; 2 - "often"; 3 - "very often." Total score for attention deficit subscale is to be formed using summations of all items. The maximum possible number of points is 27. The minimum score is 0. Higher score = more severe ADHD symptoms.
Time Frame: After 8 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 170 | 187
score on a scale
  Baseline | 18.4 (3.3) | 18.3 (3.5)
  After 4 weeks of the treatment | 15.7 (3.7) | 15.7 (3.7)
  After 8 weeks of the treatment | 13.0 (4.0) | 14.0 (4.7)
  ∆ between baseline and after 8 weeks of treatment | 5.4 (4.3) | 4.3 (4.3)
Statistical Analysis 1: Comparison: Prospekta vs Placebo; Mean changes of ADHD-RS-V scores (attention deficit subscale) after 8 weeks of treatment were compared; Test type: Superiority; p = 0.0063, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Total ADHD-RS-V Hyperactivity/Impulsivity Subscale Score
Description: Attention Deficit Hyperactivity Disorder-Rating Scale-V (ADHD-RS-V). Hyperactivity/impulsivity subscale. Versus baseline. The home version of ADHD-RS-V will be used separately for children (7-10 years old) and teenagers (11-12 years old). The home version of ADHD-RS-V includes two subscales, one for attention deficit and one for hyperactivity-impulsivity. The hyperactivity/impulsivity items are: (1) Fidgets; (2) Leaves seat; (3) Runs about; (4) Playing quietly; (5) On the go; (6) Talks excessively; (7) Blurts out answers; (8) Awaiting turns; (9) Interrupts or intrudes. Each item is responded to using a four-point Likert scale, where 0 - "never or rarely"; 1 - "sometimes"; 2 - "often"; 3 - "very often." Total score for hyperactivity/impulsivity subscale is to be formed using summations of all items. The maximum possible number of points is 27. The minimum score is 0. Higher score = more severe ADHD symptoms.
Time Frame: After 8 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 170 | 187
score on a scale
  Baseline | 14.1 (4.2) | 14.4 (4.4)
  After 4 weeks of the treatment | 11.9 (4.0) | 12.5 (4.1)
  After 8 weeks of the treatment | 9.3 (4.3) | 10.5 (4.9)
  ∆ between baseline and after 8 weeks of treatment | 4.8 (4.2) | 3.9 (4.3)
Statistical Analysis 1: Comparison: Prospekta vs Placebo; Mean changes of ADHD-RS-V scores (hyperactivity/impulsivity subscale) after 8 weeks of treatment were compared; Test type: Superiority; p = 0.0525, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: CGI-EI Efficacy Score
Description: Clinical Global Impression Efficacy Index (CGI-EI). Rating scale for assessment of the therapeutic effect of treatment and associated side effects. The scale consists of 2 items: therapeutic effect and side effects. Scores in therapeutic effect range from 1 (marked improvement) to 13 (unchanged or worse). Scores in side effects range from 0 (no side effects) to 3 (side effects outweigh therapeutic effects). Efficacy index ranges between 0 and 16. Higher values represent a worse result. CGI-EI is filled out by an investigator. It is necessary to indicate the level of efficacy of the therapy and the grade of safety of the therapy and circle the index values at the intersection of the selected lines.
Time Frame: After 8 weeks of treatment
Population: There is no data on the CGI-EI scale after 8 weeks of treatment from 4 patients in the Prospekta group and 2 patients in the Placebo group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 170 | 187
score on a scale
  Therapeutic effect | 5.9 (3.2) | 6.9 (3.1)
  Side effect | 1.0 (0.2) | 1.1 (0.3)
  Efficacy index | 6.9 (3.2) | 8.0 (3.1)
Statistical Analysis 1: Comparison: Prospekta vs Placebo; Therapeutic effect analysis; Test type: Superiority; p = 0.0024, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Prospekta vs Placebo; Side effects analysis; Test type: Superiority; p = 0.1722, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Prospekta vs Placebo; Efficacy index analysis; Test type: Superiority; p = 0.0012, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Changes in Vital Signs (Pulse Rate (Heart Rate))
Description: Based on medical records. Vital signs will be measured in a medical setting.
Time Frame: Visit 1 (Baseline), Visit 2 (4 weeks), Visit 3 (8 weeks)
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 174 | 189
beats/min
  Visit 1 | 82.9 (9.2) | 82.4 (9.5)
  Visit 2 | 83.1 (8.2) | 82.3 (8.3)
  Visit 3 | 81.9 (8.8) | 82.4 (8.1)
Statistical Analysis 1: Comparison: Prospekta vs Placebo; Test type: Superiority; p = 0.13, ANOVA — The p-value associated with "treatment*visit" interaction of changes from baseline visit 1 to visit 2 and 3 endpoint between Prospekta and Placebo treatment groups. Model includes treatment, visit and treatment*visit interaction

7. Secondary Outcome: Changes in Vital Signs (Blood Pressure)
Description: Based on medical records. Vital signs will be measured in a medical setting.
Time Frame: Visit 1 (Baseline), Visit 2 (4 weeks), Visit 3 (8 weeks)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 174 | 189
mmHg
  Systolic pressure/Visit 1 | 104.5 (9.1) | 104.0 (9.3)
  Systolic pressure/Visit 2 | 104.0 (9.0) | 103.8 (9.3)
  Systolic pressure/Visit 3 | 104.1 (9.4) | 104.1 (9.3)
  Diastolic pressure/Visit 1 | 66.9 (6.5) | 66.3 (6.3)
  Diastolic pressure/Visit 2 | 66.8 (6.3) | 66.7 (6.9)
  Diastolic pressure/Visit 3 | 66.6 (5.9) | 67.0 (6.9)
Statistical Analysis 1: Comparison: Prospekta vs Placebo; This analysis applies to Systolic pressure data; Test type: Superiority; p = 0.81, ANOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Prospekta vs Placebo; This analysis applies to Diastolic pressure data; Test type: Superiority; p = 0.22, ANOVA — [p-value comment as in outcome 6, analysis 1]

8. Secondary Outcome: Changes in Vital Signs (Respiration Rate (Breaths Per Minute))
Description: Based on medical records. Vital signs will be measured in a medical setting.
Time Frame: Visit 1 (Baseline), Visit 2 (4 weeks), Visit 3 (8 weeks)
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 174 | 189
breaths per minute
  Visit 1 | 19.9 (2.5) | 20.3 (2.8)
  Visit 2 | 20.0 (2.6) | 20.2 (2.9)
  Visit 3 | 20.1 (3.0) | 20.0 (2.7)
Statistical Analysis 1: Comparison: Prospekta vs Placebo; Test type: Superiority; p = 0.13, ANOVA — [p-value comment as in outcome 6, analysis 1]

9. Secondary Outcome: Percentage of Patients With Clinically Relevant Laboratory Abnormalities
Description: Laboratory tests include the following parameters (absolute and relative values): hematology, biochemistry and urinalysis. Laboratory tests will be made by central laboratory.
Time Frame: For 8 weeks of the treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 174 | 189
Participants | 7 | 3
Statistical Analysis 1: Comparison: Prospekta; Test type: Superiority; p = 0.2, Fisher Exact

10. Other Pre Specified Outcome: Occurrence and Type of Adverse Events (AE) During the Treatment. AE Severity.
Description: Based on medical records. AE recording is started after the first dose of the study drug (SD) and continued throughout the study therapy as well as for 24 hours after the last dose of the SD.
Time Frame: For 8 weeks of the treatment
Population: Total number of AE was 66 among 46 participants. 31 AE in 23 participants of Prospekta group, 35 AE in 23 participants of Placebo group.
Measure: Count of Units; unit: Number of AE
Units Other Than Participants: Number of AE
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 23 | 23
Number analyzed (Number of AE) | 31 | 35
Number of AE
  Light | 19 | 19
  Medium | 12 | 16
Statistical Analysis 1: Comparison: Prospekta vs Placebo; Test type: Superiority; p = 0.62, Fisher Exact

11. Other Pre Specified Outcome: Occurrence and Type of Adverse Events (AE) During the Treatment. AE Relation to the Study Drug.
Description: as for outcome 10
Time Frame: For 8 weeks of the treatment
Population: A total of 66 AEs were identified in 46 patients, including 31 AEs in 23 patients in the Prospekta group, 35 AEs in 23 participants of Placebo group.
Measure: Count of Units; unit: Number of AE
Units Other Than Participants: Number of AE
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 23 | 23
Number analyzed (Number of AE) | 31 | 35
Number of AE
  No connection | 19 | 19
  Can't be classified | 0 | 3
  Conditional | 3 | 4
  Dubious | 2 | 4
  Possible | 7 | 5
Statistical Analysis 1: Comparison: Prospekta vs Placebo; Test type: Superiority; p = 0.5, Fisher Exact

12. Other Pre Specified Outcome: Occurrence and Type of Adverse Events (AE) During the Treatment. AE Outcome.
Description: as for outcome 10
Time Frame: For 8 weeks of the treatment
Population: as for outcome 11
Measure: Count of Units; unit: Number of AE
Units Other Than Participants: Number of AE
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 23 | 23
Number analyzed (Number of AE) | 31 | 35
Number of AE
  Recovery/resolution | 25 | 20
  Recovery/resolution with consequences | 1 | 0
  No recovery/resolution | 3 | 13
  Outcome unknown | 2 | 2
Statistical Analysis 1: Comparison: Prospekta vs Placebo; Test type: Superiority; p = 0.0254, Fisher Exact

ADVERSE EVENTS:
Time Frame: During 8 weeks (start after taking the first dose of the study drug, during the entire period of the study therapy - 8 weeks and within 24 hours after the last dose of the study drug).
Arm/Group | Prospekta | Placebo
All-Cause Mortality (participants affected / at risk) | 0/174 | 0/189
Serious Adverse Events (participants affected / at risk) | 0/174 | 0/189
Other Adverse Events (participants affected / at risk) | 23/174 | 23/189
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prospekta (N=174) | Placebo (N=189)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Plaque on the tongue (Gastrointestinal disorders) | 0 (0) | 1 (1)
Belching (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — without additional clarifications
Viral infection of the respiratory tract (Infections and infestations) | 2 (2) | 6 (6)
Flu (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) — without additional clarifications
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) — without additional clarifications
Acute respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Acute nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) — without additional clarifications
Increase of white blood cells in the urine (Investigations) | 1 (1) | 0 (0)
Total cholesterol increase (Investigations) | 0 (0) | 1 (1)
AST increase (Investigations) | 1 (1) | 0 (0)
Creatinine increase (Investigations) | 1 (1) | 0 (0)
Creatinine increase in the blood (Investigations) | 2 (2) | 0 (0)
Oxalate increase in urine (Investigations) | 1 (1) | 0 (0)
Cholesterol Increase in the blood (Investigations) | 1 (1) | 0 (0)
White blood cells increase (Investigations) | 0 (0) | 1 (1)
Neutrophils increase (Investigations) | 0 (0) | 1 (1)
Shift of the leukocyte formula to the left (Investigations) | 1 (1) | 0 (0)
White blood cells decrease (Investigations) | 0 (0) | 1 (1)
Percentage of lymphocytes increase (Investigations) | 0 (0) | 1 (1)
Percentage of monocytes increase (Investigations) | 0 (0) | 1 (1)
Percentage of stab neutrophils increase (Investigations) | 0 (0) | 1 (1)
Percentage of lymphocytes decrease (Investigations) | 1 (1) | 1 (1)
Metabolic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neurodermatitis exacerbation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sweating rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3) — without additional clarifications
Tension headache (Nervous system disorders) | 0 (0) | 2 (2)
Episodic headache (Nervous system disorders) | 1 (1) | 0 (0)
Exacerbation of the present disease (General disorders) | 0 (0) | 1 (1)
General weakness (General disorders) | 1 (1) | 0 (0)
Urinary incontinence in sleep (Psychiatric disorders) | 1 (1) | 0 (0)
Obsessive-compulsive symptom (Psychiatric disorders) | 1 (1) | 0 (0)
Problems falling asleep (Psychiatric disorders) | 1 (1) | 0 (0)
Ticosis disorder, unspecified (Nervous system disorders) | 1 (1) | 0 (0)
Enuresis exacerbation (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT04569357/Prot_SAP_000.pdf